CLINICAL TRIAL: NCT03916367
Title: Clinical Outcome of CT-guided Radioactive Iodine-125 Seeds Implantation for Inoperable Early Stage Non-small Cell Lung Cancer
Brief Title: CT-guided Radioactive I-125 Seeds Implantation for Early Stage Lung Cancer
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CNRBG-81532-ESNSCLC-RISI
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-04

CONDITIONS: Early Stage Non-small Cell Lung Cancer
Keywords: radioactive iodine-125 seeds implantation; non-small cell lung cancer; early stage
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early Stage Lung Cancer: The patients with early stage non-small cell lung cancer who were treated with CT-guided radioactive iodine-125 seeds implantation during December 2010 to December 2018.
  Interventions: Radiation: CT-guided Radioactive I-125 Seeds Implantation

INTERVENTIONS:
Radiation: CT-guided Radioactive I-125 Seeds Implantation — The radioactive Iodine-125 seed can release low dose of irradiation persistently which kills tumors cell and causes less damage to normal tissue at the same time. The treatment was performed under CT monitoring.

SUMMARY:
This study observes the efficacy and side effects of CT-guided radioactive iodine-125 seed brachytherapy in inoperable early stage non-small cell lung cancer retrospectively, and analyzes the influence of clinical and dosimetric factors on the outcomes.

DETAILED DESCRIPTION:
Radioactive Iodine-125 seed brachytherapy is a conventional treatment in Peking University Third Hospital. Radioactive Iodine-125 seed brachytherapy is the implantation of Iodine-125 seed into tumors.The radioactive Iodine-125 seed can release low dose of irradiation persistently which kills tumors cell and causes less damage to normal tissue at the same time. This study collects the data of patients with early stage (stage I-II, N0) non-small cell lung cancer who underwent CT-guided radioactive Iodine-125 seed implantation from 2010 to 2018. The investigators evaluate the dose that covers 90% target volume(D90) and other parameters after the implantation. The efficacy and adverse effects were observed. Local control(LC) time and overall survival(OS) time are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* histological proven non-small cell lung cancer
* UICC (Union for International Cancer Control) stage was T1-3N0M0 (stage Ia-IIb)
* inoperable and CT-guided radioactive iodine-125 seeds brachytherapy was used as the initial treatment without external beam radiotherapy

Exclusion Criteria:

* actual dose of covers 90% target volume (D90) less than 100 Gy in postoperative validation
* case information and/or follow-up information was unavailable

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with early stage non-small cell lung cancer who were treated with CT-guided radioactive iodine-125 seeds implantation during December 2010 to December 2018 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2010-12-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Local control time | Outcomes were followed up every 3 months after enrollment. The last follow-up timepoint is February 2019.
  The time from the date of seeds implantation to the date of recurrence of the implanted tumor or the date of last observation.
Overall survival time | Outcomes were followed up every 3 months after enrollment. The last follow-up timepoint is February 2019.
  The time from the date of seeds implantation to the date of death from any cause or the date of last observation.

SECONDARY OUTCOMES:
Incidence of adverse events | Outcomes were followed up every 3 months after seeds implantation. The last follow-up timepoint is February 2019.
  The adverse events were evaluated by the common terminology criteria for adverse events (CTCAE). The rate of each adverse event was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, M.D. Ph.D., Principal Investigator — Department of Radiation Oncology, Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: CSR
Time Frame: Data will be available within 6 months of the study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.